CLINICAL TRIAL: NCT03223142
Title: A Pilot Study of Multi-mode Precision Ablation System for the Treatment of Liver Malignant
Brief Title: Standardization of Multi-modal Tumor Ablation Therapy System
Acronym: SMTATS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Fudan University (Other); Ruijin Hospital (Other); Changhai Hospital (Other); Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1604159-3-1605&1604159-3-1606
Record Dates: First submitted 2017-07-17; First posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2016-09

CONDITIONS: Liver Neoplasms; Ablation Techniques; Cryoablation; Safety; Treatment Outcome; Neoplasm Metastasis; Clinical Trial
MeSH Terms: conditions — Liver Neoplasms; Neoplasm Metastasis | interventions — Cryosurgery; Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multi-modal Precision Ablation (Experimental): In Multi-modal Precision Ablation group, patients received cryoablation immediately followed by radiofrequency ablation
  Interventions: Device: Multi-modal Precision Ablation

INTERVENTIONS:
Device: Multi-modal Precision Ablation — In Multi-modal Precision Ablation group, patients received Image-guided cryoablation immediately followed by radiofrequency ablation
  Other Names: cryoablation; radiofrequency ablation

SUMMARY:
This study will document for the safety and efficacy of image guided multi-mode precision ablation system (the combination of cryoablation and radiofrequency ablation) for the treatment of liver malignant, as well as provide the indicator of antitumor immune response for liver malignant in China.

DETAILED DESCRIPTION:
Either Cryoablation or Radiofrequency Ablation has been well accepted and widely used in clinical practice for solid tumor treatments with various commercial systems. Previous studies have established that locally exerting great thermal and mechanical stress through alternating freezing and heating abruptly broke the tumor cells and micro-vasculature in situ, enabling complete damage of primary tumor. Large amount of biological stimuli was released during this process to enhance body anti-tumor immunological response. This method thus may inhibit distal metastases and increase the survival rate. The investigators hypothesized that multi-mode thermal method (the combination of cryoablation, radiofrequency ablation) might trigger a whole body anti-tumor immune response for malignant tumor basing on multi-scale bio-thermal responses at molecular, cellular, tumor angiogenesis and tissue levels. The purpose of this study was to prospectively investigate the safety and feasibility of multi-mode precision ablation system for the treatment of liver malignant.

ELIGIBILITY:
Inclusion Criteria:

* 1.Adults aged 18 years to 70 years of either gender;
* 2. Histologically/cytologically confirmed hepatocellular carcinoma or colorectal cancer with liver metastasis, the primary lesion had underwent radical resection and without local recurrent, extrahepatic metastasis;
* 3. At least one measurable liver metastasis by RECIST criteria. No more than 5 lesions and smaller than 4.0 cm each;
* 4. Patients' liver function classified as Child-Pugh A or B, total bilirubin <=3.0 mg/dL, serum creatinine <= 2.5 mg/dL, White blood cell count >= 2.0×10^9/L, Platelets >= 100×10^9/L;
* 5. Performance Status(PS): Eastern cooperative Oncology Group (ECOG) <= 2, and life expectancy longer than three months;
* 6. Prior therapy, e.g., chemotherapy, radiation, is allowed provided that more than one month washout time is given, and recover from the previous treatment: according to the Common Terminology Criteria Adverse Events (CTC AE) version 4.0, all side effects (except for hair loss) degrading to 1 level or lower.

Exclusion Criteria:

* 1. Child-Pugh grade Class C, or tumor invasion into the portal vein;
* 2. Patient underwent previous cryoablation or other thermal ablation;
* 3. Patient underwent prior therapy, e.g., chemotherapy, radiation,or other anti-cancer medication no more than 3 weeks;
* 4. Patients with severe disorders of heart, lung, liver, kidney function or irreversible coagulation disorder;
* 5. Patients combined with other uncontrolled disease, including but not limited to: hypertension or diabetes, active infection, or mental illness or social condition that may affect the subject's compliance;
* 6. Pregnant or lactating women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-07 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Local control rate | From date of randomization until the date of progression of ablation lesion, assessed up to 5 years.
  Contrast enhanced CT or MRI was performed to evaluate Local tumor control

SECONDARY OUTCOMES:
Overall survival (OS) | From date of randomization until the date of death, assessed up to 5 years.
  Overall survival is defined as the time (in months) from the date of randomization to the death date.
Progression free survival (PFS) | From date of randomization until the date of first documented progression, recurrence or date of death from any cause, whichever came first first documented progression or date of death from any cause, whichever came first, assessed up to 5 years.
  Progression-free survival is defined as the time (in months) from the date of randomization until the date of the Investigator-assessed radiological disease progression or death due to any cause.
Complication rate | 6 months
  Number of participants with adverse events and complication

CONTACTS AND LOCATIONS:
Overall Officials: Lisaxu Xu, MD. PhD., Study Chair — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Liu P, Zhang A, Xu Y, Xu LX. Study of non-uniform nanoparticle liposome extravasation in tumour. Int J Hyperthermia. 2005 May;21(3):259-70. doi: 10.1080/02656730500068643. PMID 16019852
- [Result] Zhang A, Xu LX, Sandison GA, Cheng S. Morphological study of endothelial cells during freezing. Phys Med Biol. 2006 Dec 7;51(23):6047-60. doi: 10.1088/0031-9155/51/23/007. Epub 2006 Nov 2. PMID 17110769
- [Result] Shen Y, Liu P, Zhang A, Xu LX. Study on tumor microvasculature damage induced by alternate cooling and heating. Ann Biomed Eng. 2008 Aug;36(8):1409-19. doi: 10.1007/s10439-008-9511-2. Epub 2008 May 10. PMID 18470620
- [Result] Dong J, Liu P, Xu LX. Immunologic response induced by synergistic effect of alternating cooling and heating of breast cancer. Int J Hyperthermia. 2009 Feb;25(1):25-33. doi: 10.1080/02656730802279534. PMID 19219697
- [Result] Bai JF, Liu P, Xu LX. Recent advances in thermal treatment techniques and thermally induced immune responses against cancer. IEEE Trans Biomed Eng. 2014 May;61(5):1497-505. doi: 10.1109/TBME.2014.2314357. Epub 2014 Apr 10. PMID 24732979
- [Result] Xue T, Liu P, Zhou Y, Liu K, Yang L, Moritz RL, Yan W, Xu LX. Interleukin-6 Induced "Acute" Phenotypic Microenvironment Promotes Th1 Anti-Tumor Immunity in Cryo-Thermal Therapy Revealed By Shotgun and Parallel Reaction Monitoring Proteomics. Theranostics. 2016 Mar 21;6(6):773-94. doi: 10.7150/thno.14394. eCollection 2016. PMID 27162549